CLINICAL TRIAL: NCT02495519
Title: A Phase II Trial of Imatinib for Patients With Aggressive Desmoid Tumor (Aggressive Fibromatosis)
Brief Title: A Trial of Imatinib for Patients With Aggressive Desmoid Tumor (Aggressive Fibromatosis)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, Clinical Associate Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0074
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Fibromatosis
MeSH Terms: conditions — Fibroma | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imatinib (Experimental): Imatinib 400 mg/day until disease progression
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Imatinib 400 mg/day until disease progression

SUMMARY:
Aggressive fibromatosis (AF, also known as desmoid tumor) is a fibroproliferative neoplasm that typically arises in the abdomen but can develop at other anatomic sites, most commonly in the extremities. These tumors have a relatively high local failure rate after primary treatment using surgery and/or radiotherapy, and although rarely giving rise to distant metastases, can be multifocal and, therefore, not surgically resectable. Moreover, tumor may recur adjacent to the site of surgical resection, underscoring the limitations of surgery in the palliative setting. Therefore, effective medical therapies for AF are needed to maintain quality of life and prolong survival.The goal of the current study was to better define the activity of imatinib in the treatment of AF and to determine the molecular basis for response/nonresponse

ELIGIBILITY:
Inclusion Criteria:

1. Written consent;
2. Age ≥ 10 years;
3. Eastern Cooperative Oncology Group Performance status ≤ 2;
4. Histologically confirmed desmoid tumor;
5. Disease progression after local treatment
6. Measurable target lesion (RECIST criteria) ;
7. Adequate hematological, renal and liver functions :

Exclusion Criteria:

1. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.
2. Pregnant or lactating female
3. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
non-progressive rate | 16weeks
  non-progressive rate at 16weeks

SECONDARY OUTCOMES:
overall survival | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Song Kim, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea